CLINICAL TRIAL: NCT01018095
Title: Randomized Phase IV Trial of Metronidazole Single Dose Versus 7 Day Dose for Treatment of Trichomonas Vaginalis Among HIV-infected Women
Brief Title: Trichomonas Vaginalis Recurrence Among HIV+ Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Patricia Kissinger, Principal Investigator, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 543793; U19AI061972 (NIH)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Trichomonas Infections; HIV Infections
MeSH Terms: conditions — Trichomonas Infections; HIV Infections | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose (Active Comparator): Metronidazole 2 gm single dose
  Interventions: Drug: Metronidazole
- 7 day dose (Active Comparator): Metronidazole 500 mg dose x 7 days
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — 2 gm single dose versus 7 day 500 mg BID dose
  Other Names: Flagyl

SUMMARY:
The purpose of this study is to determine if the 2 gram single dose of metronidazole is as effective as the 7 day 500 mg BID dose for treatment of Trichomonas vaginalis (TV) among HIV-infected women.

DETAILED DESCRIPTION:
This is a Phase IV equivalency trial as both doses of metronidazole are listed in the the Centers for Disease Control and Prevention Treatment Guidelines for the treatment of T vaginalis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* HIV-positive
* TV positive by either wet preparation or culture
* ability to refrain from all alcohol use for 24 hours before and after taking oral metronidazole
* willing to take metronidazole treatment

Exclusion Criteria:

* pregnant
* incarcerated
* previously enrolled
* currently taking disulfiram
* alcoholism or known liver damage
* medical contraindications to metronidazole
* treated with metronidazole within the previous 14 days
* requires treatment for B.V. per Amsel's criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kissinger, Ph.D., Principal Investigator — Tulane University
Locations (5):
- United States (5):
  - HIV Outpatient Clinic, New Orleans, Louisiana
  - NOAIDS, New Orleans, Louisiana
  - Crossroads Clinic, Jackson, Mississippi
  - Thomas St Clinic, Houston, Texas
  - Northwest Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kissinger P, Muzny CA, Mena LA, Lillis RA, Schwebke JR, Beauchamps L, Taylor SN, Schmidt N, Myers L, Augostini P, Secor WE, Bradic M, Carlton JM, Martin DH. Single-dose versus 7-day-dose metronidazole for the treatment of trichomoniasis in women: an open-label, randomised controlled trial. Lancet Infect Dis. 2018 Nov;18(11):1251-1259. doi: 10.1016/S1473-3099(18)30423-7. Epub 2018 Oct 5. PMID 30297322
- [Derived] Kissinger P, Mena L, Levison J, Clark RA, Gatski M, Henderson H, Schmidt N, Rosenthal SL, Myers L, Martin DH. A randomized treatment trial: single versus 7-day dose of metronidazole for the treatment of Trichomonas vaginalis among HIV-infected women. J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):565-71. doi: 10.1097/QAI.0b013e3181eda955. PMID 21423852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected women undergoing a routine gynecological examination performed by a clinic health care provider between May 1, 2006 and July 17, 2009 were tested for Trichomonas Vaginalis (TV) by culture as standard of care practice in selected public HIV outpatient clinics in New Orleans, Louisiana; Houston, Texas; and Jackson, Mississippi.
Groups:
- 7 Day Dose; Single Dose: Metronidazole : 2 gm single dose versus 7 day 500 mg BID dose
Period: Overall Study
Arm/Group | 7 Day Dose | Single Dose
Started | 135 | 135
Completed | 79 | 73
Not Completed | 56 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7 Day Dose | Single Dose | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 135 | 134 | 269
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (9.3) | 40.7 (9.4) | 40.1 (9.4)
Gender [Count of Participants; unit: Participants]
  Female | 135 | 135 | 270
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 135 | 135 | 270

OUTCOME MEASURES:

1. Primary Outcome: TV Culture Positive Result
Description: At the participants' test of cure (TOC) visits they were screened for Trichomonas vaginalis using (InPouch) culture. Presence of parasite will yield a culture positive result.
Time Frame: test-of-cure visit at 6-12 days post-treatment completion
Population: Participants who returned for their test of cure visit
Measure: Number; unit: participants
Arm/Group | 7 Day Dose | Single Dose
Number analyzed (Participants) | 130 | 125
participants | 11 | 21
Statistical Analysis 1: Comparison: 7 Day Dose vs Single Dose; It was initially estimated that a total of 380 participants (190 per arm) would be required, with 90% power and a significance level of 5%, to establish equivalency between the two treatment arms.31 Enrollment rates were lower than estimated and only 270 participants (135 per arm) were enrolled; Test type: Non-Inferiority or Equivalence — Continuous variables were assessed for normality, and tested accordingly. When appropriate, continuous variables were categorized using clinically relevant cut-points. Categorical variables were compared using the Chi-square test. The measure of association at TOC was calculated as a relative risk with 95% confidence interval; p = .045, Relative risk; The measure of association at TOC and 3 months was calculated as a relative risk with 95% confidence interval; Risk Ratio (RR) = 0.5, 95% CI 2-sided [0.25 to 1.00], Standard Error of Mean 0.191
Statistical Analysis 2: Comparison: 7 Day Dose vs Single Dose; Test type: Non-Inferiority or Equivalence — It was initially estimated that a total of 380 participants (190 per arm) would be required, with 90% power and a significance level of 5%, to establish equivalency between the two treatment arms; p < 0.05, Chi-squared — Continuous variables were assessed for normality, and tested accordingly. When appropriate, continuous variables were categorized using clinically relevant cut-points. Categorical variables were compared using the Chi-square test; Risk Ratio (RR) = 0.46, 95% CI 2-sided [0.21 to 0.98], Standard Deviation 1

2. Secondary Outcome: TV Culture Positive Result
Description: Participants who returned for their follow up visits were tested for Trichomonas vaginalis using InPouch culture. If parasites are present, it will yield a culture positive result.
Time Frame: 3 months post-enrollment
Population: Participants who returned for their 3 mo follow up visit
Measure: Number; unit: participants
Arm/Group | 7 Day Dose | Single Dose
Number analyzed (Participants) | 73 | 79
participants | 8 [7.3 to 14.7] | 19 [19.3 to 28.9]
Statistical Analysis 1: Comparison: 7 Day Dose vs Single Dose; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Continuous variables were assessed for normality, and tested accordingly. When appropriate, continuous variables were categorized using clinically relevant cut-points. Categorical variables were compared using the Chi-square test. The measure of association at 3 months was calculated as a relative risk with 95% confidence interval; p = 0.03, Relative risk; The measure of association at TOC and 3 months was calculated as a relative risk with 95% confidence interval; Risk Ratio (RR) = 0.46, 95% CI 2-sided [.21 to 0.98], Standard Error of Mean 0.196

ADVERSE EVENTS:
Time Frame: 4 years and 2 months
Arm/Group | 7 Day Dose | Single Dose
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/135
Other Adverse Events (participants affected / at risk) | 0/135 | 0/135

LIMITATIONS AND CAVEATS:
Generalizability is always a concern in clinical trials, however our findings are likely generalizable to the majority of HIV-infected women in the U.S. though studies in Caucasian and Hispanic women are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No